CLINICAL TRIAL: NCT04660929
Title: A Phase 1, First in Human Study of Adenovirally Transduced Autologous Macrophages Engineered to Contain an Anti-HER2 Chimeric Antigen Receptor in Subjects With HER2 Overexpressing Solid Tumors
Brief Title: CAR-macrophages for the Treatment of HER2 Overexpressing Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Carisma Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 101
Record Dates: First submitted 2020-11-23; First posted 2020-12-09 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-04

CONDITIONS: HER2-positive; Adenocarcinoma; Bile Duct Cancer; Biliary Tract Cancer; Bladder Cancer; Breast Cancer; Breast Neoplasm; Carcinoma, Ductal; Carcinoma, Hepatocellular; Cancer; Lung Cancer, Non-Small-Cell; Carcinoma, Ovarian Epithelial; Carcinoma, Small Cell; Carcinoma, Squamous; Carcinoma, Transitional Cell; Colorectal Cancer; Esophagogastric Junction Neoplasms; Inflammatory Breast Cancer; Stomach Neoplasms; Malignant Neoplasms; Ovarian Neoplasms; Pancreatic Cancer; HER2-positive Solid Tumors; HER2-positive Breast Cancer; HER2-positive Gastric Cancer; HER-2 Protein Overexpression; HER-2 Gene Amplification; Prostate Cancer; Head and Neck Cancer; Endometrial Cancer; Lung Cancer, Small Cell
Keywords: HER2-positive solid tumors; Phase 1; cell therapy; CAR-macrophage; immunotherapy; advanced cancer; post menopausal; premenopausal; metastatic cancer; Prostate Cancer; Head and Neck Cancer; Lung Cancer, Small Cell; Endometrial Cancer; Lung Cancer, Non-Small Cell
MeSH Terms: conditions — Adenocarcinoma; Bile Duct Neoplasms; Biliary Tract Neoplasms; Urinary Bladder Neoplasms; Breast Neoplasms; Carcinoma, Ductal; Carcinoma, Hepatocellular; Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Ovarian Epithelial; Carcinoma, Small Cell; Carcinoma, Squamous Cell; Carcinoma, Transitional Cell; Colorectal Neoplasms; Inflammatory Breast Neoplasms; Stomach Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms; Prostatic Neoplasms; Head and Neck Neoplasms; Endometrial Neoplasms; Small Cell Lung Carcinoma; Neoplasm Metastasis | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 and Group 2 (Experimental): Both groups will receive the full dose manufactured per patient. Group 1 will undergo intra subject dose escalation of IV administrations of up to 500 million total cells on Day 1, up to 1.5 billion total cells on Day 3, and up to 3.0 billion total cells on Day 5. Group 2 will receive the full dose IV on Day 1 of up to 5 billion cells total.
  Interventions: Biological: CT-0508
- Intraperitoneal Administration (Experimental): All cohorts will receive the full dose manufactured per patient. Cohorts 1-3 will undergo intrasubject dose escalations of IP administration as follows:
  Cohort 1 up to 500 million total cells on Day 1, up to 1 billion total cells on Day 3 and up to 1.5 billion total cells on Day 5.
  Cohort 2 up to 1.5 billion total cells on Day 1, up to 2 billion total cells on Day 3 and any remaining cells on Day 5.
  Cohort 3 up to 2.5 billion total cells on Day 1 and up to 2.5 billion total cells on Day 3.
  Cohort 4 will 1 dose on Day 1 of up to 5 billion total cells.
  Interventions: Biological: CT-0508
- 89[Zr]radiolabeled CT-0508 (Experimental): 89[Zr] radiolabeled group will receive a full dose IV on Day 1 of up to 500 million total cells of 89[Zr] radiolabeled CT-0508 and non-radiolabeled CT-0508 of up to 4.5 billion total cells (Univ of Penn Abramson Cancer Center only).
  Interventions: Biological: CT-0508
- CT-0508 in Combination with Pembrolizumab (Experimental): All regimen levels will receive the full dose manufactured per patient up to 5 billion total cells. Regimen Levels 1 and 2 will undergo intrasubject dose escalations of IV administration as follows:
  Regimen Level 1: up to 500 million total cells on Day 1, up to 1.5 billion total cells on Day 3, and up to 3.0 billion total cells on Day 5 plus pembrolizumab 200 mg q3w starting on Day 8.
  Regimen Level 2: up to 500 million total cells on Day 1, up to 1.5 billion total cells on Day 3, and up to 3.0 billion total cells on Day 5 plus pembrolizumab 200 mg q3w starting on Day 1.
  Regimen Level 3 will receive the full dose IV on Day 1 of up to 5 billion total cells plus pembrolizumab 200 mg q3w starting on Day 1.
  Interventions: Biological: CT-0508; Biological: Pembrolizumab

INTERVENTIONS:
Biological: CT-0508 — anti-HER2 CAR macrophages
Biological: Pembrolizumab — anti-PD antibody
  Other Names: Keytruda
  Arms: CT-0508 in Combination with Pembrolizumab

SUMMARY:
Phase 1, first-in-human, open label study of CAR macrophages in HER2 overexpressing solid tumors.

DETAILED DESCRIPTION:
A Phase 1, First in Human Study of Adenovirally Transduced Autologous Macrophages Engineered to Contain an Anti-HER2 Chimeric Antigen Receptor in Subjects with HER2 Overexpressing Solid Tumors

Main Study - Group 1 and Group 2 all HER2 overexpressing solid tumors

Intraperitoneal Substudy - HER2 overexpressing peritoneal disease

89[Zr] radiolabeled CT-0508 Substudy - All HER2 overexpressing solid tumors (Univ of Penn, Abramson Cancer Center only)

CT-0508 Combination with Pembrolizumab Substudy - All HER2 overexpressing solid tumors

ELIGIBILITY:
Inclusion Criteria:

* HER2-positive recurrent or metastatic solid tumors for which there are no available curative treatment options.

  * Breast cancer and gastric/gastroesophageal junction cancers must have failed approved HER2-targeted agents.
  * Other HER2-positive tumor types must have failed standard of care therapies, while prior therapy with anti-HER2 drugs is not required.
* Subject must be willing and able to undergo tumor tissue biopsy procedures
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Subject has adequate bone marrow and organ function

Exclusion Criteria:

* HIV, active hepatitis B or hepatitis C infection.
* Diagnosis of immunodeficiency or chronic exposure to systemic corticosteroid therapy or any other form of immunosuppressive therapy
* Untreated or symptomatic central nervous system (CNS) metastases or cytology proven carcinomatous meningitis.

  o Subjects with small, asymptomatic CNS metastases that do not require treatment are permitted to enroll.
* Left ventricular ejection fraction (LVEF) <50% as determined by ECHO or multiple gated acquisition scan (MUGA)

Other protocol-defined Inclusion/Exclusion may apply.

CT-0508 in Combination with Pembrolizumab Substudy Only:

Exclusion Criteria:

* Subjects with severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients
* Subjects with an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs).
* Subjects who have a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Subjects who have had an allogeneic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-02-02 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Assess the safety and tolerability of CT-0508 by estimating the frequency and severity of adverse events in subjects with HER2 overexpressing solid tumors. | 14 months
  Frequency and severity of adverse events including, but not limited to, estimating frequency and severity of Cytokine Release Syndrome (CRS)
Assess the feasibility of manufacturing CT-0508 by describing the percentage of products passing release criteria. | 12 months
  Percentage of products that pass release criteria among all manufactured products.
Assess the safety and tolerability of CT-0508 in combination with pembrolizumab by estimating the frequency and severity of adverse events in subjects with HER2 overexpressing solid tumors (CT-0508 and pembrolizumab substudy only) | 14 months
  Frequency and severity of adverse events including, but not limited to, estimating frequency and severity of Cytokine Release Syndrome (CRS)

SECONDARY OUTCOMES:
Estimate the objective response rate (ORR), according to RECIST v1.1, of at least 1 dose of CT-0508 among subjects with HER2 overexpressing solid tumors. | 24 months
  Proportion of subjects with an objective response (either a complete response [CR] or partial response [PR]) in subjects who received at least 1 dose of CT-0508 and at least the 8-week tumor evaluation as determined by the investigator using RECIST v1.1.
Estimate progression-free survival (PFS). | 24 months
  Defined as the time between the date of first dose and the date of first documented disease progression as determined by the investigator using RECIST v1.1 or death due to any cause, whichever occurs first.
  Defined as the time between the date of first dose and the date of first documented disease progression as determined by the investigator using RECIST v1.1 or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Jeanett Wetzel, Study Director — Carisma Therapeutics
Locations (7):
- United States (7):
  - City of Hope National Medical Center, Duarte, California
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - OHSU Knight Cancer Institute, Portland, Oregon
  - Abramson Cancer Center, Philadelphia, Pennsylvania
  - Tennessee Oncology / Sarah Cannon Research Institute, Nashville, Tennessee
  - M D Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klichinsky M, Ruella M, Shestova O, Lu XM, Best A, Zeeman M, Schmierer M, Gabrusiewicz K, Anderson NR, Petty NE, Cummins KD, Shen F, Shan X, Veliz K, Blouch K, Yashiro-Ohtani Y, Kenderian SS, Kim MY, O'Connor RS, Wallace SR, Kozlowski MS, Marchione DM, Shestov M, Garcia BA, June CH, Gill S. Human chimeric antigen receptor macrophages for cancer immunotherapy. Nat Biotechnol. 2020 Aug;38(8):947-953. doi: 10.1038/s41587-020-0462-y. Epub 2020 Mar 23. PMID 32361713
- [Derived] Reiss KA, Angelos MG, Dees EC, Yuan Y, Ueno NT, Pohlmann PR, Johnson ML, Chao J, Shestova O, Serody JS, Schmierer M, Kremp M, Ball M, Qureshi R, Schott BH, Sonawane P, DeLong SC, Christiano M, Swaby RF, Abramson S, Locke K, Barton D, Kennedy E, Gill S, Cushing D, Klichinsky M, Condamine T, Abdou Y. CAR-macrophage therapy for HER2-overexpressing advanced solid tumors: a phase 1 trial. Nat Med. 2025 Apr;31(4):1171-1182. doi: 10.1038/s41591-025-03495-z. Epub 2025 Feb 7. PMID 39920391
- [Derived] Sly LM, McKay DM. Macrophage immunotherapy: overcoming impediments to realize promise. Trends Immunol. 2022 Dec;43(12):959-968. doi: 10.1016/j.it.2022.10.002. Epub 2022 Oct 29. PMID 36441083